CLINICAL TRIAL: NCT06364878
Title: New Non-invasive Cellular and Molecular Diagnostics of Microbial Keratitis
Brief Title: Non-invasive Diagnostics of Microbial Keratitis
Status: Recruiting | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: 813533
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-04

CONDITIONS: Infectious Keratitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Tear film on Schirmers test stored in microtubes at -80°C for biochemical analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patents with suspected infectious keratitis
  Interventions: Diagnostic Test: In vivo confocal microscopy; Diagnostic Test: Tear film sampling
- Healthy controls
  Interventions: Diagnostic Test: In vivo confocal microscopy; Diagnostic Test: Tear film sampling

INTERVENTIONS:
Diagnostic Test: In vivo confocal microscopy — The patients cornea will be examined non-invasively by IVCM
  Other Names: IVCM
Diagnostic Test: Tear film sampling — Patients tear film will be collected and stored at -80 degrees for analysis

SUMMARY:
Infectious keratitis is a significant cause of partial vision loss and blindness and places a large burden on eye care professionals. One of the main challenges for the ophthalmologist when presented with a case of suspected microbial keratitis is the determination of the subtype of keratitis. It must be determined whether the origin of the infection is bacterial, viral, fungal, or parasitic, in order to prescribe a correct, effective treatment aimed at the causative pathogen. In daily practice this can be challenging, and general treatments with antibiotics are prescribed. Some cases then experiences deterioration, resulting in more patients visits and further rounds of invasive treatments and progressive vision deterioration.

This project is designed to break this cycle of nonspecific diagnosis, suboptimal treatment, and progressive worsening of vision with increased interventions. New, advanced diagnostics will be brought into the clinic to provide additional information which, if our hypothesis is correct, will result in more rapid and accurate diagnosis of the keratitis subtype. This will translate into earlier administration of a more targeted treatment, avoiding the repeated round of non-targeted treatment and progressive worsening of the patient's vision. This can directly reduce to number of clinic visits and specialist time required for treatment and follow-up of keratitis, knowledge of how the eye responds to various microbes by initiating a specific cascade of molecular inflammatory signals and changes in protein expression in the tear film.

Using in vivo confocal microscopy (IVCM) we will document the cellular status of the cornea and identify microbes infecting the cornea in real-time. Secondly, tear samples will be obtained from patients with keratitis to evaluate and quantify the molecular cytokine signatures associated with specific microbial species, confirmed by microbiological culture. We will for the first time develop cytokine profiles for the various types of infection, identifying diagnostic cytokines which in the longer term can lead to development of rapid point-of-care biomarker diagnostics.

The project aims are translated into the following hypotheses:

H1: In vivo confocal microscopy imaging features detect microbial keratitis consistent with clinical assessment and outcome at a greater frequency than microbiological culture results.

H2: Cytokine profiles (or a subset of molecules) in the eye are specific for viral, bacterial, fungal, or amoebic keratitis; and H3: A combination of in vivo confocal microscopy and molecular profiling of the tear film can yield a specific keratitis diagnosis closely matching the clinical progression and outcome of keratitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected infectious keratitis in patients over 18 years of age
* Patients with acceptable travel distance to the hospital
* Patients accepting to be part of the study

Exclusion Criteria:

* Previously diagnosed infectious keratitis during the last 6 months
* Over 50 percent thinning of the cornea
* Previous use of antibiotics (other than Chloramphenicol)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with clinically suspected infectious keratitis, over 18 years of age, presenting to the ophthalmology department at Arendal hospital.
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2028-04-08 (Estimated)

PRIMARY OUTCOMES:
IVCM findings and cytokine profile in infectious keratitis is specific for the different microbial subtypes. | 18 months
  A combination of in vivo confocal microscopy and molecular profiling of the tear film can yield a specific keratitis diagnosis closely matching the clinical progression and outcome of keratitis.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Lagali, Principal Investigator — Sorlandet Hospital HF
Locations (1):
- Sorlandet hospital, Arendal, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Currently there is not a plan to share individual data outside the project group due to confidentiality. If the investigators later would want to do this, new applications to the correct boards are needed.